CLINICAL TRIAL: NCT03033043
Title: A Prospective, Multicenter, Non-Blinded, Non-Randomized Study of the RelayPro Thoracic Stent-Graft in Subjects With an Acute, Complicated Type B Aortic Dissection
Brief Title: Study of the RelayPro Thoracic Stent-Graft in Subjects With an Acute, Complicated Type B Aortic Dissection
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bolton Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IP-0017-16
Record Dates: First submitted 2017-01-24; First posted 2017-01-26 (Estimated); Last update posted 2025-11-06 (Actual); Status verified 2025-09

CONDITIONS: Aortic Dissection Type B
Keywords: aortic; dissection; type B; thoracic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Experimental: Relay Pro (Experimental): The Relay Pro arm includes subjects who receive the device. The Relay Pro Stent Graft System is administered to treat complicated Type B aortic dissections.
  Interventions: Device: Relay Pro Stent-Graft

INTERVENTIONS:
Device: Relay Pro Stent-Graft — Endovascular treatment of an aortic dissection
  Other Names: Relay Pro Stent Graft System

SUMMARY:
This clinical trial is a prospective, multicenter, non-blinded, non-randomized study designed to assess the RelayPro thoracic endografts in the treatment of acute, complicated type B aortic dissection. The primary endpoint will measure all-cause mortality at 30 days post-procedure.

DETAILED DESCRIPTION:
This clinical trial is a prospective, multicenter, non-blinded, non-randomized study designed to assess the RelayPro thoracic endografts in the treatment of acute, complicated type B aortic dissection. The primary endpoint will measure all-cause mortality at 30 days post-procedure.

Subjects will be enrolled on a first come, first serve basis; however, no single investigational site may enroll more than 20% of the proposed sample size of up to 80 subjects. A subject is considered enrolled when arterial access is gained and an attempt is made to introduce the RelayPro Thoracic Stent-Graft. Enrollment is expected to begin in mid-2016 and complete by the end of 2020.

All subjects enrolled, as defined above, will be included in the patient population for the primary safety analyses. All subjects implanted with the RelayPro Thoracic Stent-Graft will be included in the patient population for the primary effectiveness analyses.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have an acute (symptom onset to diagnosis within 2 weeks)or subacute, complicated type B aortic dissection (entire dissection is distal to the left subclavian artery (LSA)), confirmed by Computed Tomography Angiography (CTA) or Magnetic Resonance Angiogram (MRA), with time from symptom onset to diagnosis ≤ 6 weeks, with at least one of the following:

  * Malperfusion of the viscera, kidneys, spinal cord, or lower extremities, measured by clinical or radiographic evidence;
  * Rupture;
  * Intractable pain.
* Proximal and distal aortic neck with diameter between 19 mm and 42 mm.
* Subject's anatomy must meet all of the following anatomical criteria:

  1. Proximal attachment zone distal to the left common carotid and a distal attachment zone proximal to the origin of the celiac artery. (Dissection is permitted in the distal attachment zone but is not permitted in the proximal attachment zone.)
  2. The length of the attachment zones will depend on the intended stent-graft diameter and type of graft selected.
  3. The proximal attachment zone should be 15 mm for 22 - 28 mm RelayPro grafts with bare stent (20 mm for RelayPro grafts with non-bare stent), 20 mm for 30 - 46 mm RelayPro grafts with bare stent (25 mm for RelayPro grafts with non-bare stent), and proximal to non-dissected segment (healthy zone).
  4. The distal attachment zone should be 20 mm for all RelayPro grafts.
  5. Coverage of the left subclavian artery is permitted with mandatory revascularization if patent left internal mammary artery (LIMA) bypass or left upper extremity (LUE) arteriovenous graft or anomalous vertebral artery off the aorta. Revascularization must be performed prior to device placement, and may occur during implant procedure, provided it is before coverage of the LSA by the endograft.
* Proximal attachment zone containing a straight segment (non-tapered, non-reverse-tapered, defined by <10% diameter change) with lengths equal to or greater than the required attachment length for the intended device.
* Vascular dimensions (e.g., aortic diameters, length from left subclavian to celiac artery) must be in the range that can be safely treated with the RelayPro Thoracic Stent-Grafts.
* Adequate iliac or femoral artery access for introduction of the RelayPro Delivery System. Alternative methods to gain proper access may be utilized (e.g., iliac conduit).
* Subject willing to comply with the follow-up evaluation schedule.
* Subject (or Legally Authorized Representative, LAR) agrees to sign an Informed Consent Form prior to treatment.

Exclusion Criteria:

* Diagnosis of traumatic injury or transection of the descending thoracic aorta.
* Significant stenosis, calcification, thrombus, or tortuosity of intended fixation sites that would compromise fixation or seal of the device.
* Planned coverage of left carotid or celiac arteries; or anatomic variants that would compromise circulation to the carotid, vertebral, or innominate arteries after device placement, which is not amenable to subclavian revascularization.
* Prior endovascular or surgical repair in the descending thoracic aorta. The device may not be placed within any prior endovascular or surgical graft.
* Concomitant aneurysm/disease of the ascending aorta, aortic arch, or abdominal aorta, requiring repair. Dissection extension into the abdominal aorta is acceptable.
* Prior abdominal aortic aneurysm repair (endovascular or surgical) that was performed less than 6 months prior to the planned stent implant procedure.
* Major surgical or medical procedure within 30 days prior to the planned procedure, or is scheduled for a major surgical or medical procedure within 30 days post implantation. This excludes any planned procedures for the prospective stent-graft placement.
* Untreatable allergy or sensitivity to contrast media or device components, including metal stents.
* Known or suspected connective tissue disorder.
* Blood coagulation disorder or bleeding diathesis for which the treatment cannot be suspended for one week pre- and/or post-repair.
* Coronary artery disease with unstable angina.
* Severe congestive heart failure (New York Heart Association functional class IV).
* Stroke and/or Myocardial Infarction (MI) within 3 months of the planned treatment date.
* Pulmonary disease requiring the routine (daily or nightly) need for oxygen therapy outside the hospital setting.
* Acute renal failure or chronic renal insufficiency, and not receiving dialysis.
* Hemodynamically unstable.
* Active systemic infection and/or mycotic aneurysms.
* Bowel necrosis.
* Morbid obesity or other condition that may compromise or prevent the necessary imaging requirements.
* ASA risk classification = V (Moribund patient not expected to live 24 hours with or without operation).
* Less than two-year life expectancy.
* Current or planned participation in an investigational drug or device study that has not completed primary endpoint evaluation.
* Currently pregnant or planning to become pregnant during the course of the study.
* Medical, social, or psychological issues that Investigator believes may interfere with treatment or follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality post-procedure | 30 days
  All-cause mortality 30 days post-procedure

SECONDARY OUTCOMES:
Technical Success at the time of the index procedure | During deployment of the device
  Successful delivery and deployment of the device, including withdrawal of the delivery system;
Treatment success through 1 month | 1 month, 6 months, 12 months, and annually through 5 years, defined as individual endpoints and as a composite
  * Absence of Major adverse Event (MAE)
  * Absence of relevant MAEs:
  * Paraplegia;
  * Paraparesis;
  * New ischemia due to branch vessel compromise;
  * Absence of unintentional rupture of the dissection septum;
Dissection Treatment Success | 1, 6, and 12 month follow-up visits, and annually through 5 years.
  • Dissection treatment success through 1 month, 6 months, 12 months, and annually through 5 years, defined as individual endpoints and as a composite

CONTACTS AND LOCATIONS:
Overall Officials: Christian Shults, MD, Principal Investigator — Medstar Health Research Institute; Peter Rossi, MD, Principal Investigator — Medical College of WI
Locations (21):
- United States (21):
  - USC Department of Surgery, Los Angeles, California
  - University of Colorado Denver, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Yale School of Medicine, New Haven, Connecticut
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - St. Vincent Heart Center, Indianapolis, Indiana
  - University of Iowa Hospital and Clinic, Iowa City, Iowa
  - University of Maryland Medical Center (UMB), Baltimore, Maryland
  - University of Michigan Health System, Ann Arbor, Michigan
  - Buffalo General Medical Center, Buffalo, New York
  - University Hospitals, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Providence Heart Institute, Portland, Oregon
  - University of Pennsylvania Medical Center / Penn Presbyterian, Philadelphia, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Sentara Heart Hospital, Norfolk, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - University of Washington, Seattle, Washington
  - Medical College of WI, Vascular Surgery, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No